CLINICAL TRIAL: NCT06619834
Title: Pilot Trial of Financial Navigation and Peer Support to Improve Diabetes Outcomes
Brief Title: Financial Navigation and Peer Support to Improve Diabetes Outcomes
Acronym: FNaPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Minal Patel, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HUM00243207
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Navigation only (Active Comparator): Financial navigation using software called TailorMed only. The professional Financial Navigator is from the TailorMed team.
  Interventions: Behavioral: Financial Navigation Only
- Financial Navigation and Peer Support (Active Comparator): Financial navigation using software called TailorMed combined with peer support. The professional Financial Navigator is from the TailorMed team. Peer Supporters will be trained community members recruited from Michigan Medicine.
  Interventions: Behavioral: Financial Navigation and Peer Support

INTERVENTIONS:
Behavioral: Financial Navigation and Peer Support — A combined intervention of technology-supported financial navigation and peer support: A professional financial navigator from TailorMed will use the software to assist participants in exploring options to reduce their specific economic barriers to treatment and care, and non-medical social risks. Participants will also be matched with a Peer Supporter to help improve the participants' diabetes self-management.
  Arms: Financial Navigation and Peer Support
Behavioral: Financial Navigation Only — A professional financial navigator from TailorMed will use the software to assist participants in exploring options to reduce their specific economic barriers to treatment and care, and non-medical social risks.
  Arms: Financial Navigation only

SUMMARY:
The goal of this clinical trial pilot study is to test the feasibility, acceptability, and preliminary efficacy of a combined intervention strategy of 1) technology-supported financial navigation to address economic burden of disease and 2) peer support both to facilitate linkages to clinical care and community resources to address social risks and improve participants' diabetes self-management. The main aims of this pilot study are:

* To examine the feasibility and acceptability of technology-supported financial navigation and financial navigation with peer support
* To examine trends in preliminary efficacy of technology-supported financial navigation and peer support versus financial navigation-alone on 1) A1c and blood pressure (primary outcomes), and 2) out-of-pocket costs, treatment-related financial stress, cost-related non-adherence behaviors, diabetes distress, diabetes self-care behaviors, and uptake of social care assistance (secondary outcomes).

The investigators will assess whether a combined intervention of technology-supported financial navigation and peer support will produce trends in superior diabetes and social care outcomes to financial navigation alone via a 2-arm randomized controlled trial.

Participants will

* Complete 3 survey appointments at baseline, and 3 and 6 months. Each appointment will consist of a survey assessment, an HbA1C test, and two blood pressure readings over the phone.
* Be randomized to either financial navigation only or financial navigation and peer support.

ELIGIBILITY:
Inclusion Criteria:

Participants:

* 18-75 years of age
* diagnosis of diabetes with prescribed anti-hyperglycemic medication
* most recent (within the past 6 months) recorded hemoglobin A1c (HbA1c) level of ≥7.5% for individuals ≤70 years and >8.0% for individuals between 70-75 years in age
* positive report of financial burden or cost-related non-adherence (CRN) using screening questions developed and validated from prior work 20-22
* be willing to provide personal health information in order to effectively participate in the intervention

Peer Supporters:

* International Classification of Diseases (ICD)-10 code for diabetes
* In the past had A1cs' > 8.0% but whose most recent A1c in the prior 12 months is <8.0%.
* Past experience with economic burden or unmet social risk factors
* Adults 18-75 years

Exclusion Criteria:

Participants:

* a diagnosis of a serious psychiatric disorder (e.g., schizophrenia)
* active alcohol or illicit drug use
* current pregnancy or planning pregnancy
* taking a medication that alters glucose metabolism (e.g., oral steroids)
* report a comorbidity expected to limit life span to < 3 years
* Participation in another diabetes study, but the investigators will ask them if they would like to be peer supporters

Peer Supporters:

* A diagnosis of a serious psychiatric disorder (e.g., schizophrenia)
* Active alcohol or illicit drug use
* Current pregnancy or planning pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
A1c | From enrollment to the end of participant study duration at 6 months
  Collect A1c sample using A1c Now SelfCheck test kit
Blood Pressure | From enrollment to the end of participant study duration at 6 months
  Measure participant blood pressure using the Omron home blood pressure monitor. Both systolic and diastolic blood pressure will be measured.

SECONDARY OUTCOMES:
Uptake of social care assistance | From enrollment to the end of participant study duration at 6 months
  Adapted from Your Current Life Situation (YCLS) and Health Leads Screening Tools
Successfully having social/financial need address | From enrollment to the end of participant study duration at 6 months
  Enrollment data from TailorMed software
Cost-related non-adherence behaviors | From enrollment to the end of participant study duration at 6 months
  Individual survey items adapted from National Health Interview Survey (NHIS)
Out-of-pocket costs | From enrollment to the end of participant study duration at 6 months
  Data generated from TailorMed software
Diabetes-related social support | From enrollment to the end of participant study duration at 6 months
  Diabetes Support Scale (DSS) Minimum value- Strongly Disagree, Maximum value- Strongly Agree Higher score mean a better outcome.
Diabetes self-care behaviors | From enrollment to the end of participant study duration at 6 months
  Diabetes Self-care Activities Scale - Adapted Minimum value- 0 Days, Maximum value- 7 Days Higher scores mean a better outcome.
Social needs screening | From enrollment to the end of participant study duration at 6 months
  Accountable Health Communities Health-Related Social Needs Screening Tool (Q15-17) and Item adapted from National Health Interview Survey (Q18)
  Adapted from Accountable Health Communities Health-Related Social Needs Screening Tool, Health Leads Social Needs Screening Toolkit, & Kaiser Permanente Your Current Life Situation Questionnaire
  Minimum value- Never True, Maximum value- Often True. Higher scores mean worse outcome.
Diabetes Distress | From enrollment to the end of participant study duration at 6 months
  Diabetes Distress Scale (DDS2 version)
  Minimum Value- Not a Problem, Maximum Value- Serious Problem Higher scores mean worse outcome.
Treatment-related financial stress | From enrollment to the end of participant study duration at 6 months
  COmprehensive Score for financial Toxicity (COST)-Functional Assessment of Chronic Illness Therapy (FACIT) domains adapted for diabetes
  The score includes reverse-coding 6-items, summing all items, multiplying sum by 11 and dividing the total by number of items answered. Lower scores indicate higher perceptions of financial burden. (Min value of 0, max value of 44)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underlie results in a publication, after de-identification.
Supporting Information: SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: The data will be made available to other researchers who provide a methodologically sound proposal and who have appropriate approvals from all relevant Institutional Review Boards (IRBs). The data will be shared for analyses to achieve aims in the approved proposal. Data will be shared through a secure File Transfer Protocol (FTP) site through encryption protocols that allow secure uploading of files with data sharing limited to specific users. Select datasets will also be made available through the University of Michigan openICPSR Repository (http://www.icpsr.umich.edu/icpsrweb/deposit/index.jsp). Proposals should be directed to minalrp@umich.edu. To gain access, data requestors will need to sign a data access agreement.